CLINICAL TRIAL: NCT03841149
Title: Measurement of Kidney Volume and Renal Tumor Volume Using 3D-Ultrasound Imaging
Brief Title: Volume 3D_US Kidney
Acronym: VolUS3D
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI18037J; 2018-A01394-51 (Other: N° ID-RCB)
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Diseases; Renal Tumor
Keywords: 3D Ultrasound volume measurements; Renal volume; Tumour Volume
MeSH Terms: conditions — Renal Insufficiency, Chronic; Carcinoma, Renal Cell | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- VolUS3D patients: Patients with renal tumour
  Interventions: Other: Ultrasound Imaging

INTERVENTIONS:
Other: Ultrasound Imaging — 3D volume calculation using on-line and off-line softwares
  Other Names: 3D Ultrasound transducer and fusion imaging

SUMMARY:
The purpose of this study is to measure the volume of the kidney and tumors using 3D-US acquisition and to correlate these measurements to contrast-enhanced CT or MRI.

DETAILED DESCRIPTION:
Additional objectives are comparison between true volume measurements and volume estimation using measurements of the three perpendicular diameters, comparison of inter and intra variability of 3D US measurements with inter and intra variability of 3D CT or MRI measurements, calculation of 3D and 2D volume measurements during contrast-enhanced US examination when the injection is performed for clinical routine purposes such as vascular and extension staging, during interventional procedures such as US guided biopsy targeting the non-necrotic tumour parenchyma. Concordance between 2D and 3D US acquisitions will be compared to CT and MRI measurements. Comparison of volume measurements between non-contrast and contrast-enhanced methods (US, CT and MRI) will be performed. The results will be compared to renal function before and after tumour treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age 18)
* Absence of participant's opposition
* No contra-indication to contrast-enhanced CT AND MRI (a single contrast-enhanced imaging modality is sufficient)
* Affiliated to Social Security

Exclusion Criteria:

- Contra-indication to both contrast-enhanced CT AND MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (n=80) referred for renal tumour management (including imaging, biopsy or percutaneous ablation)
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
3D-US volume measurements | 1 month
  Kidney and renal tumor

SECONDARY OUTCOMES:
2D-US volume measurements | 1 month
  Kidney and renal tumor
Inter and intra variability measurements | 1 month
  Kidney and renal tumor
2D and 3D US volume measurements during Contrast-enhanced US (if performed for patient management) | 1 month
  Kidney and renal tumor

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Correas, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No